CLINICAL TRIAL: NCT00270218
Title: A Phase I Clinical Trial to Evaluate Immune Response Kinetics and Safety of Two Different Primes, Adenoviral Vector Vaccine (VRC-HIVADV014-00-VP) and DNA Vaccine (VRC-HIVDNA009-00-VP), Each Followed by Adenoviral Vector Boost in Healthy, HIV-1 Uninfected Adults
Brief Title: Safety of and Immune Response to Two Different HIV Vaccines, Each Followed by a Adenoviral Vaccine Boost, in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 068; 10060 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2005-12-21; First posted 2005-12-26 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Adenoviral Vector Vaccine; DNA Plasmid Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 1 (Experimental): Arm 1 participants will be given an injection of VRC-HIVADV014-00-VP vaccine on Days 0 and 168.
  Interventions: Biological: VRC-HIVADV014-00-VP
- 2 (Placebo Comparator): Arm 2 participants will be given an injection of final formulation buffer (FFB) on Days 0 and 168.
  Interventions: Biological: FFB
- 3 (Experimental): Arm 3 participants will be given an injection of VRC-HIVDNA009-00-VP vaccine on Days 0 and 28. Participants will also be given an injection of VRC-HIVADV014-00-VP on Day 168.
  Interventions: Biological: VRC-HIVADV014-00-VP; Biological: VRC-HIVDNA009-00-VP
- 4 (Placebo Comparator): Arm 4 participants will be given an injection of phosphate buffered saline (PBS) on Days 0 and 28 and an injection of FFB on Day 168.
  Interventions: Biological: FFB; Biological: PBS

INTERVENTIONS:
Biological: VRC-HIVADV014-00-VP — HIV-1 recombinant adenoviral vector vaccine given as a 1 mL intramuscular injection in the deltoid
  Arms: 1; 3
Biological: VRC-HIVDNA009-00-VP — HIV-1 DNA plasmid vaccine given as a 1 mL intramuscular injection in the deltoid
  Arms: 3
Biological: FFB — Adenoviral vector FFB given as a 1 mL intramuscular injection in the deltoid
  Arms: 2; 4
Biological: PBS — phosphate buffered saline
  Arms: 4

SUMMARY:
The purpose of this study is to determine the safety of and immune response to an adenoviral vector HIV vaccine or a DNA HIV vaccine, each followed by an adenoviral vector HIV vaccine boost, in HIV uninfected adults.

DETAILED DESCRIPTION:
Evaluating the immunogenicity of HIV vaccines is critical to improving vaccine design and development. The adenoviral vector HIV vaccine VRC-HIVADV014-00-VP has shown immunogenicity in early studies and appeared safe and well tolerated at three different doses in a prior dose-escalation vaccine trial in HIV uninfected adults. The DNA HIV vaccine VRC-HIVDNA009-00-VP has shown immunogenicity in multiple clinical trials; in one trial, the DNA vaccine demonstrated a nearly 100% CD4 T-cell response rate. The DNA plasmids in both vaccines code for proteins from HIV subtypes A, B, and C, which together represent 90% of new HIV infections. This study will determine the safety and immune response to the administration of an adenoviral vector HIV vaccine or a DNA HIV vaccine, each followed by an adenoviral vaccine boost, in HIV uninfected adults.

This study will last 1 year. Participants will be randomly assigned to one of two groups. Within each group, participants will be randomly assigned to receive either vaccine or control injections. Group 1 participants will receive either placebo or the adenoviral HIV vaccine at study entry and Month 6. Group 2 participants will receive either placebo or the DNA HIV vaccine at study entry and Month 1 and the adenoviral HIV vaccine at Month 6. Participants will be asked to record their temperatures and other side effects in a symptom log on the day of each vaccination and for 3 days thereafter to report any side effects.

Group 1 participants will have 16 study visits, and a physical exam and HIV and pregnancy prevention counseling will occur at each visit. Participants will also be asked about any side effects and medications they are taking. Blood collection will occur at most visits. Urine collection will occur at selected visits. Participants will be asked to complete a social impact assessment at Months 2, 6, and 12 and a testing and belief questionnaire at Months 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Good general health
* Pre-existing adenovirus 5 (Ad5) neutralizing antibody titers of less than a 1:12 ratio
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (anti-HCV) antibody negative or negative HCV PCR if anti-HCV antibody is positive
* Have access to a participating HIV Vaccine Trials Unit (HVTU) and are willing to be followed during the study
* Willing to receive HIV test results
* Understand the vaccination procedure
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV trial. Participants who can provide documentation that they received a placebo in a prior HIV trial may be eligible.
* Immunosuppressive medications within 168 days prior to first study vaccination
* Blood products within 120 days prior to first study vaccination
* Live attenuated vaccines within 30 days prior to first study vaccination
* Investigational research agents within 30 days prior to first study vaccination
* Medically indicated subunit or killed vaccines within 14 days prior to first study vaccination
* Current anti-tuberculosis (TB) preventive therapy or treatment
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health. More information about this criterion can be found in the protocol.
* Any medical, psychiatric, or social condition that would interfere with the study. More information about this criterion can be found in the protocol.
* Any job-related responsibility that would interfere with the study
* Serious adverse reactions to vaccines, including hypersensitivity and related symptoms. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection. Participants who have been fully treated for syphilis for more than 6 months prior to study entry are not excluded.
* Moderate to severe asthma. More information on this criterion can be found in the protocol.
* Type 1 or type 2 diabetes mellitus. Participants with histories of isolated gestational diabetes are not excluded.
* Thyroid disease or surgical removal of the thyroid requiring medication during the 12 months prior to study entry
* Accumulation of fluid in the blood vessels (angioedema) within 3 years prior to study entry if episodes are considered serious or have required medication in the 2 years prior to study entry
* Uncontrolled hypertension
* Body mass index (BMI) of 40 or greater OR BMI of 35 or greater if certain other criteria apply. More information about these criteria can be found in the protocol.
* Bleeding disorder
* Cancer. Participants with surgically removed cancer that is unlikely to recur are not excluded.
* Seizure disorder
* Absence of the spleen
* Mental illness that would interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2006-02; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity signs and symptoms, laboratory measures, and adverse and serious experiences) | After each injection and for 6 months after the last injection
Magnitude of HIV-specific CD4+ and CD8+ T-cell responses, defined as percentage of T cells expressing IFN-gamma or IL-2 to vaccine peptide pools | Within first 6 weeks following primary adenoviral vaccination, the second DNA vaccination, and the booster adenoviral vaccination
Social impact (negative experiences or problems associated with participation in the study and other social, travel, work, school, health care, life insurance, health insurance, housing, military, or other impacts identified by the participant) | Throughout the study

SECONDARY OUTCOMES:
Expression of HIV-specific T-cell memory differentiation markers and other markers of interest by flow cytometry | Within first 6 weeks following primary adenoviral vaccination, the second DNA vaccination, and the booster adenoviral vaccination
Titer to HIV-specific binding antibodies assessed by ELISA | Within first 6 weeks following primary adenoviral vaccination, the second DNA vaccination, and the booster adenoviral vaccination
Titer of HIV-specific neutralization antibodies assessed by neutralizing antibody assay, if indicated | Within first 6 weeks following primary adenoviral vaccination, the second DNA vaccination, and the booster adenoviral vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Stephen De Rosa, MD, Study Chair — Fred Hutchinson Cancer Research Center and University of Washington; Spyros A. Kalams, MD, Study Chair — Vanderbilt University
Locations (7):
- United States (7):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - NY Blood Ctr./Union Square CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Background] Barouch DH, Nabel GJ. Adenovirus vector-based vaccines for human immunodeficiency virus type 1. Hum Gene Ther. 2005 Feb;16(2):149-56. doi: 10.1089/hum.2005.16.149. PMID 15761255
- [Background] De Rosa SC, Lu FX, Yu J, Perfetto SP, Falloon J, Moser S, Evans TG, Koup R, Miller CJ, Roederer M. Vaccination in humans generates broad T cell cytokine responses. J Immunol. 2004 Nov 1;173(9):5372-80. doi: 10.4049/jimmunol.173.9.5372. PMID 15494483
- [Background] Shiver JW, Emini EA. Recent advances in the development of HIV-1 vaccines using replication-incompetent adenovirus vectors. Annu Rev Med. 2004;55:355-72. doi: 10.1146/annurev.med.55.091902.104344. PMID 14746526
- [Background] Vanniasinkam T, Ertl HC. Adenoviral gene delivery for HIV-1 vaccination. Curr Gene Ther. 2005 Apr;5(2):203-12. doi: 10.2174/1566523053544236. PMID 15853728
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067